CLINICAL TRIAL: NCT00047879
Title: A Phase II Study of Peg-Interferon Alpha-2B (Peg-Intron(TM)) and Thalidomide in Adults With Recurrent High-Grade Gliomas
Brief Title: Phase II Trial of Peginterferon Alpha-2b and Thalidomide in Adults With Recurrent Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Howard A. Fine, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030002; 03-C-0002 (Other: Clinical Center (CC), National Institutes of Health (NIH)); 030002 (Other: Clinical Center (CC), National Institutes of Health (NIH)); NCT00052650 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2002-10-23 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-09

CONDITIONS: Glioma
Keywords: Brain Tumors; Experimental; Toxicities; Efficacy; Progression-Free; Brain Tumor; Glioma
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — peginterferon alfa-2b; peginterferon alfa-2a; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glioblastoma multiforme stratum (Other): Glioblastoma multiforme is one of the most common and aggressive types of brain tumor.
  Interventions: Biological: PEG-interferon alfa-2b; Drug: Thalidomide
- Anaplastic Glioma Stratum (Other): Anaplastic glioma is a type of brain tumor that develops from star-shaped glial cells that support nerve cells. Anaplastic oligodendroglioma is a malignant type of brain tumor sensitive to treatment with chemotherapy and radiotherapy.
  Interventions: Biological: PEG-interferon alfa-2b; Drug: Thalidomide

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — 0.3 µg/kg of IFN alfa-2b (PEG-Intron once weekly) plus daily oral thalidomide, subcutaneous injection
  Other Names: Pegasys
Drug: Thalidomide — Two 50mg tablets (100 mg total dose) every night before bedtime starting on day one.
  Other Names: Thalomid

SUMMARY:
This study will examine the safety and effectiveness of peginterferon alpha-2b (PEG-Intron) alone and together with thalidomide in patients with gliomas (a type of brain tumor). Gliomas are nourished by blood delivered through blood vessels whose formation is stimulated by substances produced by the tumor itself. Stopping the growth of new vessels can slow or prevent tumor growth. The Food and Drug Administration has approved various interferons for treating several diseases, including melanoma and some leukemias. These drugs block new vessel growth in patients with recurrent tumors, but in high doses they produce serious side effects. Therefore, this study will use a low dose of PEG-Intron given weekly instead of high doses given several times a week. Thalidomide, currently approved to treat leprosy, also blocks development of new blood vessel formation. In a recent study of thalidomide given to 36 patients with gliomas, 4 patients had tumor shrinkage, 12 had stable disease for at least 2 months, and at least 3 had responses to treatment lasting 6 to 14 months.

Patients 18 years of age and older with a primary glioma whose tumor has recurred or is growing following standard treatment and does not respond to radiation therapy may be eligible for this study. Candidates will be screened with a physical examination, blood and urine tests (including a pregnancy test for women of childbearing potential), and magnetic resonance imaging (MRI) or computed tomography (CT) of the head.

Patients will continue treatment cycles as long as the drug is tolerated without serious side effects and the tumor is not growing. While on the study, patients will undergo various tests and procedures as follows:

Physical and neurologic examinations every 6 weeks MRI or CT brain scan every 6 weeks to assess tumor status. MRI is a diagnostic test that uses a strong magnetic field and radio waves to show structural and chemical changes in tissues. During the scan, the patient lies on a table in a narrow cylinder containing a magnetic field. He or she can speak with a staff member through an intercom system at all times during the procedure.

DETAILED DESCRIPTION:
Background:

There is a growing belief that angiogenesis inhibition represents a potentially promising, novel therapeutic approach to highly vascular solid tumors like malignant gliomas. Thalidomide and Peg-Intron (IFN - Interferon) are attractive drugs to use in combination to test the hypothesis of combination anti-angiogenesis therapy inhibition given their proven activity as single agents in patients with malignant gliomas and their spectrum of largely non-overlapping toxicities.

Given recent preclinical data describing more potent antiangiogenic and anti-tumor effects of low dose, continuous IFN administration, we are interested in evaluating the use of pegylated IFN in combination with thalidomide. Thus, we are proposing a phase II trial of pegylated IFN with thalidomide in patients with recurrent gliomas.

Objectives:

To obtain preliminary evidence of anti-tumor efficacy of PEG-Intron in combination with thalidomide in patients with recurrent high grade gliomas as assessed by prolongation of progression-free survival compared to historical controls.

A secondary endpoint in this trial is to determine the response rate associated with the combination therapy in each of the two strata and to evaluate and document all toxicities from PEG-Intron in combination with thalidomide at the doses prescribed in this protocol in this patient population.

Eligibility:

Patients with histologically proven supratentorial malignant primary gliomas will be eligible for this protocol. These include glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified).

Patients must not have received prior therapy with Peg-Intron or Thalidomide.

Design:

Patients will be treated with weekly PEG-Intron plus daily oral thalidomide. All patients will be treated for 6 weeks following which patients will have a repeat MRI scan to assess disease response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven supratentorial malignant primary gliomas will be eligible for this protocol. These include glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified).
* Patients must have evaluable or measurable disease and have shown unequivocal evidence for tumor recurrence or progression by MRI or CT scan. This scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and the initiation of treatment, a new 20 baseline MR/CT scan is required. The same type of scan, i.e., MRI or CT must be used throughout the period of treatment for tumor measurement.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as the following conditions apply:
* They have recovered from the effects of surgery
* Measurable disease following resection of recurrent tumor is not mandated for eligibility into the study. Patients must have evaluable disease.
* To best assess the extent of residual disease post-operatively, a CT/MRI should be done no later than 96 hours in the immediate post-operative period or 4-6 weeks post-operatively. If the 96 hour scan is more than 2 weeks from registration, the scan needs to be repeated.
* The baseline on-study MR/CT is performed within 14 days of registration and on a steroid dosage that has been stable. If the steroid dose is increased between the date of imaging and the initiation of Peg-Intron with or without Thalidomide, a new baseline MR/CT is required on stable steroids for 5 days.
* Patient must have failed prior radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, MR spectroscopy or surgical documentation of disease.
* Prior therapy. There are no limitations to number of prior therapies.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be > 18 years old, and with a life expectancy > 8 weeks.
* Patients must have a Karnofsky performance status of > 60.
* Patients must have recovered from the toxic effects of prior therapy (including resolution of effects on laboratory values): 2 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy, 2 weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents e.g. tamoxifen, cis- retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the PI.
* Patients must have adequate bone marrow function (WBC > 3,000/l, ANC > 1,500 mm3, platelet count of > 100,000/mm3, and hemoglobin > 10 gm%), adequate liver function (SGOT and bilirubin < 2 times the upper limit of normal), and adequate renal function (creatinine < 1.5 mg/dL or creatinine clearance > 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.
* Patients must not be pregnant or nursing, and all patients (both men and women) must be willing to practice birth control for 1 month prior, during and for 4 months after treatment with thalidomide. It has been proposed that thalidomide may interfere with hormonal-based contraception, therefore, barrier methods of contraception (i.e. diaphragm, condom) MUST be used rather than, or in addition to birth control pills.
* No peripheral neuropathy > grade 1.
* No concurrent use of other investigational agents.

Exclusion Criteria:

* Patients must not have:
* Serious active infection
* Disease that will obscure toxicity or dangerously alter drug metabolism
* Serious intercurrent medical illness.
* Significant illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy.
* Patients must not have received prior therapy with Peg-Intron or Thalidomide.
* Concurrent chemotherapy, immunotherapy, or radiotherapy is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Fine, M.D., Principal Investigator — NCI, NIH
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dinapoli RP, Brown LD, Arusell RM, Earle JD, O'Fallon JR, Buckner JC, Scheithauer BW, Krook JE, Tschetter LK, Maier JA, et al. Phase III comparative evaluation of PCNU and carmustine combined with radiation therapy for high-grade glioma. J Clin Oncol. 1993 Jul;11(7):1316-21. doi: 10.1200/JCO.1993.11.7.1316. PMID 8315428
- [Background] Takamiya Y, Friedlander RM, Brem H, Malick A, Martuza RL. Inhibition of angiogenesis and growth of human nerve-sheath tumors by AGM-1470. J Neurosurg. 1993 Mar;78(3):470-6. doi: 10.3171/jns.1993.78.3.0470. PMID 8433151
- [Background] Fine HA, Figg WD, Jaeckle K, Wen PY, Kyritsis AP, Loeffler JS, Levin VA, Black PM, Kaplan R, Pluda JM, Yung WK. Phase II trial of the antiangiogenic agent thalidomide in patients with recurrent high-grade gliomas. J Clin Oncol. 2000 Feb;18(4):708-15. doi: 10.1200/JCO.2000.18.4.708. PMID 10673511
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus
- See also: Drug Information Portal — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We planned to accrue 32 patients to the GBM stratum and 32 patients to the AG stratum.
  The accrual ceiling was 64 patients on this trial. We anticipated accruing these patients within one year of opening this study.
Period: Overall Study
Arm/Group | Glioblastoma Multiforme Stratum | Anaplastic Glioma Stratum
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Progressive disease | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glioblastoma Multiforme Stratum | Anaplastic Glioma Stratum | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.85) | 53.67 (11.93) | 54.71 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival is defined as the percent of patients that are progression free and alive 6 months after initiating therapy.
  Progression of disease by > 50% increase in the size of the tumor compared to baseline after the first cycle only, and then >25% increase in the size of the tumor for all subsequent cycles.
Time Frame: 6 months
Population: The primary objective was not met. Only registered 7 out of 64 participants and they all came off the study for progressive disease around 3-4 months after starting the study. None of the participants were evaluated for progression-free survival at 6 months because the study was stopped at 4 months due to progressive disease.
Measure: Number; unit: Percent of participants
Arm/Group | Glioblastoma Multiforme Stratum | Anaplastic Glioma Stratum
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Complete or Partial Response
Description: Response is defined per RECIST criteria. Measurable disease is defined as bidimensionally measurable lesions with clearly defined margins by CT or MRI scan.
  Evaluable disease is defined as unidimensionally measurable lesions, masses with margins not clearly defined, or lesions with a multiple cystic component.
  Complete response (CR) is complete disappearance of all measurable and evaluable disease. Partial response (PR) is greater than or equal to 50% decrease under baseline in the sum of products or perpendicular diameters of all measurable lesions.
Time Frame: 6 months
Population: Registered 7 out of 64 participants and they came off study for progressive disease around 3-4 months after starting the study.
Measure: Number; unit: Participants
Arm/Group | Glioblastoma Multiforme Stratum | Anaplastic Glioma Stratum
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 4 months
Measure: Number; unit: Participants
Arm/Group | Glioblastoma Multiforme Stratum | Anaplastic Glioma Stratum
Number analyzed (Participants) | 4 | 3
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Glioblastoma Multiforme Stratum | Anaplastic Glioma Stratum
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glioblastoma Multiforme Stratum (N=4) | Anaplastic Glioma Stratum (N=3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Metabolic, hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Elevated AST (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glioblastoma Multiforme Stratum (N=4) | Anaplastic Glioma Stratum (N=3)
edema: limb right upper extremity (General disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Metabolic, ALT elevated (Investigations) | 1 (1) | 0 (0)
Pain, skin (Nervous system disorders) | 1 (1) | 0 (0)
Mood alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
AST (Investigations) | 1 (1) | 0 (0)
Glucose (Investigations) | 1 (1) | 0 (0)
Elevated AST (Investigations) | 1 (1) | 0 (0)
Elevated bilirubin (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neurology, somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, other leg/foot cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Registered 7 out of 64 participants and they came off study for progressive disease around 3-4 months after starting the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No